CLINICAL TRIAL: NCT00037102
Title: An Open Label Study of the Safety and Efficacy of Combination Therapy With AVONEX and Bi-Monthly High Dose Intravenous Methotrexate With Leucovorin Rescue in the Treatment of Multiple Sclerosis
Brief Title: Combination Therapy With Avonex and BiMonthly High Dose Intravenous Methotrexate in Multiple Sclerosis
Acronym: MTX01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MidAmerica Neuroscience Research Foundation at Rowe Neurology Institute (Other)
Collaborators: Consultants in Neurology (Industry); Biogen (Industry)
Responsible Party: Principal Investigator, Vernon D. Rowe III, MD, Vernon D. Rowe III, MD, MidAmerica Neuroscience Research Foundation at Rowe Neurology Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MANI-MTX01-001
Record Dates: First submitted 2002-05-15; First posted 2002-05-17 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing; Methotrexate; AVONEX; interferon beta 1a; demyelinating; autoimmune
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — Interferon beta-1a; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: interferon beta 1a
Drug: methotrexate

SUMMARY:
The participant will receive weekly intramuscular treatment with AVONEX® (interferon beta 1-a) and bi-monthly high dose intravenous methotrexate with Leucovorin rescue.

DETAILED DESCRIPTION:
The participant will receive weekly intramuscular treatment with AVONEX® (interferon beta 1-a) and bi-monthly high dose intravenous methotrexate with Leucovorin rescue. Entrance into the study will be based on Multiple Sclerosis Functional Composite Score (MSFC) evaluations at -4 months, and - 1 month prior to study, where a decrease in score is noted. The composite score consists of the Timed 25-Foot Walk, Nine-Hole Peg Test (9HPT), and Paced Auditory Serial Addition Test 3 (PASAT 3). The patient must have been on AVONEX® for at least 6 months.

At study entrance, baseline lab work (complete blood count, platelet count, routine electrolytes, blood urea nitrogen, creatinine, liver function tests, 24 hour urine collection for creatinine clearance, and urine pH), an electrocardiogram (measurement of heart activity) and serum pregnancy test will be done. A complete physical examination will be performed, including measurements of vital signs (heart rate and blood pressure), as well as magnetic resonance imaging (MRI) to document status of disease. A self-administered questionnaire, the MSQLI (Multiple Sclerosis Quality of Life Instrument), will be completed at baseline and at the end of the study. MSFC and safety evaluations (previously mentioned blood and urine tests and electrocardiograms (EKG), will be conducted throughout the study at months 2, 4, 6, 8, 10, and 12. Blood tests of immune cells will also be drawn at these visits. The patient can continue this regimen of treatment at their own discretion and cost, and outside the parameters of this study, if there is apparent efficacy without serious adverse events. This treatment would be under the supervision of Dr. Rowe.

The patients will continue their AVONEX® intramuscular injections of 30 micrograms (administered by patient or caregiver) on a weekly basis with scheduled intravenous high dose methotrexate at 2 Gm/m2 followed by intravenous and oral leucovorin rescue once every 2 months. The methotrexate infusions will be performed in our outpatient infusion center. The patient will be required to complete a patient diary during the course of the trial, participate in and keep all scheduled appointments, and to inform the research staff and physician of any change in concomitant medications or adverse events that they may experience.

ELIGIBILITY:
To be eligible for entry into this study, candidates must meet the following eligibility criteria at the time of enrollment:

* Between the ages of 18 and 60 years, inclusive.
* Diagnosis of clinically definite relapsing MS.
* Must have been on AVONEX® therapy for at least six months.
* Brain MRI scans demonstrating lesions consistent with MS.
* Subject must have had at least one clinical exacerbation in the last year, and this must have occurred after having been on AVONEX® therapy for at least six to twelve (6-12) months. A clinical exacerbation is defined as a decrease of 0.1 in the MSFC composite or any of the subset domains scores administered 3 months apart.
* Give written informed consent prior to any testing under this protocol, including screening tests and evaluation that are not considered part of the subject's routine care.

To be eligible for treatment with methotrexate, subjects must have evidence for MS disease activity on their baseline screening MRI.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2001-07; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vernon D ROWE, MD, Principal Investigator — MidAmerica Research Foundation